CLINICAL TRIAL: NCT00961948
Title: A Pilot Study for the Determination of Inter-observer Variation for Abnormalities Detected by Indigo Carmine Staining and Narrow Band Imaging Among Patients Undergoing Surveillance Colonoscopy for Ulcerative Colitis
Brief Title: Indigo Carmine Staining and Narrow Band Imaging (NBI) of Colonic Mucosa for Detection of Dysplasia in Ulcerative Colitis
Status: Completed | Type: Observational
Sponsor: Mayo Clinic (Other)
Responsible Party: Michael F. Picco, M..D., Mayo Clinic Florida
Other Study IDs: 09-000196
Record Dates: First submitted 2009-08-18; First posted 2009-08-19 (Estimated); Last update posted 2013-02-27 (Estimated); Status verified 2013-02

CONDITIONS: Ulcerative Colitis
Keywords: Indigo carmine dye spraying; Narrow band imaging (NBI); Confocal Microscopy
MeSH Terms: conditions — Colitis, Ulcerative

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

SUMMARY:
A prospective, randomized trial to determine indigo carmine dye spraying and narrow band imaging (NBI) of colonic mucosa to detect dysplasia in ulcerative colitis (UC). Confocal laser microscopy may be beneficial in the further assessment of abnormalities identified by these methods.

DETAILED DESCRIPTION:
Specific Aims:

Primary:

1. To assess intra- and inter-observer agreement for the detection of abnormalities seen by white light colonoscopy followed by indigo carmine staining and white light colonoscopy followed by NBI imaging.

   Secondary:
2. To estimate the sensitivity and specificity of these modalities for dysplasia among UC patients who undergo surveillance colonoscopy.
3. To assess intra- and inter-observer agreement for abnormalities identified by confocal laser microscopy among patients with chronic ulcerative colitis.
4. To determine the specificity and sensitivity of confocal microscopy in the detection of dysplasia among patients with ulcerative colitis.

50 consecutive patients with clinically quiescent UC presenting for surveillance colonoscopy will be randomized to white light followed by NBI OR white light followed by indigo carmine staining. Identified abnormalities will then be targeted for confocal imaging in 40 patients. Immediately prior to confocal imaging, fluorescein 2.5 ml of 10% solution will be administered intravenously. For these patients, confocal images will also be obtained of the area around the lesion and of the colon segments as in the parent study and correlated with pathology. Gross activity will be determined by white light colonoscopy for each colon segment. At least 32 biopsies for surveillance will be obtained with additional biopsies of abnormalities present on white light, NBI or indigo carmine. Photographs will be obtained of all abnormalities prior to biopsy and of random mucosa without abnormalities. Intra- and inter-observer agreement will be based on the first 10 patients at each site through review of de-identified endoscopic photographs. If modifications are necessary because of poor agreement, re-assessment will be made after the next 10 patients. Otherwise each site will enroll 40 additional patients with agreement summarized and sensitivity and specificity of these techniques for detecting dysplasia

Significance: If intra and inter-observer agreement for mucosal abnormalities detected by indigo carmine and NBI modalities is shown to be good, in ulcerative colitis, then larger studies will be planned on UC surveillance populations. If confocal techniques are feasible then these will be integrated into larger studies.

ELIGIBILITY:
Inclusion Criteria:

1. Clinically quiescent (UC) disease will be defined as a colitis activity index <8 at the time of enrollment.
2. Scheduled for routine, clinically-indicated colonoscopy surveillance

Exclusion Criteria:

1. Patients unable to give informed consent,
2. Pregnant or female patients of child bearing age who are sexually active an not practicing birth control methods. (in this group a pregnancy test is required as per routine clinical care)
3. Poor colonic preparation (<90% colon visualization)
4. Documented allergy to indigo carmine
5. Coagulopathy that can not be corrected (INR> 1.5 and/or platelet count<50,000)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with clinically quiescent, histologically proven pan-ulcerative colitis for at least 8 years will be recruited from the outpatient gastroenterology clinic of the Mayo Clinic Florida and randomized to white light followed by NBI or white light followed by indigo carmine staining to include confocal microscopy.
Sampling Method: Probability Sample
Enrollment: 60 (Actual)
Dates: Start 2009-06; Primary Completion 2013-02 (Actual); Study Completion 2013-02 (Actual)

PRIMARY OUTCOMES:
Overall estimates of inter- and intra-observer positive and negative agreement of at least 80% for the detection of abnormalities seen by white light colonoscopy followed by indigo carmine staining and white light colonoscopy followed by NBI imaging. | two years

SECONDARY OUTCOMES:
Confocal laser microscopy may be beneficial in the further assessment of abnormalities identified by these methods of white light colonoscopy followed by indigo carmine staining and white light colonoscopy followed by NBI imaging. | two years

CONTACTS AND LOCATIONS:
Overall Officials: Michael F Picco, M.D., Principal Investigator — Mayo Clinic
Locations (1):
- Mayo Clinic Florida, Jacksonville, Florida, United States